CLINICAL TRIAL: NCT04495075
Title: The Use of Visuomotor Therapy to Modulate Corticospinal Excitability in Patients Following ACL-Reconstruction
Brief Title: Neuromuscular Control in Individuals Following ACL-Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Joseph Hart, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20441
Record Dates: First submitted 2020-07-21; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Anterior Cruciate Ligament Injuries; Quadriceps Muscle Atrophy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: Laboratory Controlled Crossover Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessing investigator was blinded to the intervention that was received by the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visuomotor Therapy (Experimental): Patients were seated in the isokinetic dynamometer with their hips flexed to 85º. A target sine wave with a maximum amplitude of 30% MVIC and a minimum amplitude of 5% MVIC and a frequency of 0.128 Hz was visually presented to the patient.31 The patient was instructed to match their torque to the presented target throughout the duration of testing. Each visuomotor therapy trial was 60-seconds, followed by 30-seconds of rest for 10 repetitions, totaling 15 minutes.
  Interventions: Other: Visuomotor Therapy
- Passive Motion (Active Comparator): Patients were seated in the isokinetic dynamometer with their hips flexed to 85º. The dynamometer then passively moved the patient from 80º to 120º of knee flexion for 60-seconds, followed by 30-seconds of rest for 10 repetitions, totaling 15 minutes. The patient was provided visual feedback of their knee position throughout the trials. The patient was instructed to relax their knee throughout the intervention.
  Interventions: Other: Passive Motion

INTERVENTIONS:
Other: Visuomotor Therapy — The use of visual feedback informing internal physiological processes, such as muscle activation, torque, and joint position, has been termed "visuomotor therapy". Visuomotor therapy encompasses completion of sub-maximal motor control tasks accompanying real-time visual biofeedback.
  Other Names: Motor Biofeedback
  Arms: Visuomotor Therapy
Other: Passive Motion — The knee is passively moved through a range of motion.
  Arms: Passive Motion

SUMMARY:
The purpose of this study is to investigate the neurophysiological contributors to muscle function following ACL Reconstruction and the influence of motor control biofeedback exercise on measures of muscle function. The research team hypothesizes that the application of motor biofeedback will increase cortical excitability of the quadriceps compared to the passive movement of the knee.

This is a single session cross-over intervention study with a 1-week washout period between treatment arms.

DETAILED DESCRIPTION:
1. Pre-treatment neuromuscular assessment Cortical Active Motor Threshed We will measure motor evoked potentials with the use of a Transcranial magnetic stimulator (MagStim model 200, Magstim Co., Ltd., Wales, UK). The MagStim has FDA 510K Clearance for stimulation of peripheral nerves.

   * The participant will be asked to sit in the dynamometer (Biodex, System 3) in knee extension at 90 degrees of knee flexion.
   * EMG electrodes will be placed on the distal quadriceps

     o Local shaving, debridement, and cleaning will be done prior if necessary
   * A non-latex swim cap will be placed on the participants head for investigator's measurements
   * Briefly, a magnetic field with a maximum value of 2.2 Tesla will be introduced to the scalp at a location in the pre-motor cortex that corresponds to the quadriceps. Single pulse stimulations will be delivered with no less than 10 seconds between stimulations (maximum = 0.1 Hz).
   * When the magnetic field is received at the premotor cortex at the appropriate area, a motor signal is sent to the quadriceps. We will record this signal with surface EMG electrodes that are on the quadriceps.
   * The participant will be asked to extend their leg to match a force equivalent to 5% MVIC. Feedback will be provided to the participant to provide such force.
   * Stimulation of the TMS will happen once every ten seconds until the Active Motor Threshold was found by the investigator.

     * The motor evoked potential measured by the quadriceps will be recorded at 80%, 90%, 100%, 110%, 120%, 130%, 140%, and 150% of the patients Active motor threshold.
2. Patient randomization

   - The patient is then randomized to 1 of 2 treatment arms. 1) Visuomotor Therapy or 2) Passive Motion
3. Perform Randomized Treatment Visuomotor Therapy

   * The participant will sit in the Biodex chair with the tested limb secured in the dynamometer
   * The participant will receive live real-time biofeedback of their knee force output (no more than 30% of maximum force)
   * The participant will aim to match their force output to a target threshold presented on the screen.
   * The participant will complete 10 60-second trials of this exercise with a 30 second rest between each trial.

   OR

   Passive Motion
   * The participant will sit in the Biodex chair with the tested limb secured in the dynamometer
   * The dynamometer will passively move the patients lower limb between 80 to 120 degrees of knee flexion
   * The participant will be asked to relax for the duration of testing - The participant will complete 10 60-second trials of this exercise with a 30 second rest between each trial.
4. Reassess Neuromuscular outcome (Step 1)
5. 1-week washout period
6. Repeat Steps 1 through 4 but the patient receives the cross-over arm intervention

ELIGIBILITY:
Inclusion Criteria:

* • Ages 18-45

  * At the time point of return to play progression following ACL Reconstruction
  * Physically active individuals based on current ACSM guidelines of 30 minutes of moderate-intensity daily physical activity three days a week)

Exclusion Criteria:

* Subjects who are known to be pregnant (self-reported)

  * Subjects diagnosed with malignancy
  * Subjects with serious infection near the lower limb
  * Subjects with known muscular abnormalities
  * History of cardiopulmonary disorder
  * Subjects with a previous history of stroke
  * History of neurological or psychiatric disorders including poorly controlled migraine headaches, seizure disorder, history or immediate family history of seizures and/or epilepsy
  * Subjects with any type of neuropathy (numbness and tingling)
  * Subjects with a clinical diagnosis of multiple sclerosis (MS) or Parkinson's Disease
  * Implanted biomedical device (active or inactive implants (including device leads), including deep brain stimulators, cochlear implants, and vagus nerve stimulators)
  * History of skull fracture
  * Subjects who have any metal implants anywhere in their head, neck or shoulders
  * Patients taking any medications, which may influence cortical excitability, which could influence neurophysiologic measures) and affect objective clinical data (e.g. antispastics, anxiolytics, hypnotics, ant-epileptics)
  * Subjects who are prescribed medications which may influence cortical excitability, which could influence neurophysiologic measures) and affect objective clinical data (e.g. antispastics, anxiolytics, hypnotics, ant-epileptics), will not be able to remain in the study.
  * Unable to provide consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps Motor Evoked Potential (micoVolts) PreSham (Passive Motion) | 6-months post-Anterior Cruciate Ligament Reconstruction
  Activation of the Quadriceps muscle through stimulation of primary motor cortex. Measured Through electromyography on the vastus medialis
Quadriceps Motor Evoked Potential (micoVolts) PostSham (Passive Motion) | 6-months post-Anterior Cruciate Ligament Reconstruction
  Activation of the Quadriceps muscle through stimulation of primary motor cortex. Measured Through electromyography on the vastus medialis
Change in Quadriceps Motor Evoked Potential - Sham (Passive Motion) | 6-months post-Anterior Cruciate Ligament Reconstruction
  Difference in microVolts between pre-sham measure and post-sham measure
Quadriceps Motor Evoked Potential (micoVolts) PreActive (Visuomotor Therapy) | 6-months post-Anterior Cruciate Ligament Reconstruction
  Activation of the Quadriceps muscle through stimulation of primary motor cortex. Measured Through electromyography on the vastus medialis
Quadriceps Motor Evoked Potential (micoVolts) PostActive (Visuomotor Therapy) | 6-months post-Anterior Cruciate Ligament Reconstruction
  Activation of the Quadriceps muscle through stimulation of primary motor cortex. Measured Through electromyography on the vastus medialis
Change in Quadriceps Motor Evoked Potential - Active (Visuomotor Therapy) | 6-months post-Anterior Cruciate Ligament Reconstruction
  Difference in microVolts between pre-active measure and post-active measure

CONTACTS AND LOCATIONS:
Overall Officials: Joe M Hart, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No